CLINICAL TRIAL: NCT05608460
Title: Pediatric Cervical Spine Clearance: A Multicenter Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Katie Russell, MD, Principal Investigator, University of Utah
Other Study IDs: C-Spine
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cervical Spine Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective multicenter observational study, led by Dr. Katie Russell of Intermountain Primary Children's Hospital, that will examine the sensitivity, specificity, negative, and positive predictive values of CT scan and plain films in diagnosing cervical spine injury that requires treatment. This study is funded by the Primary Children's Hospital foundation.

ELIGIBILITY:
Inclusion Criteria:

* Any participant less than 18 years old after blunt trauma
* Seen by trauma service
* With cervical spine imaging (XR, CT, or MRI)

Exclusion Criteria:

* CT scan from outside facility is poor quality and not repeated (<63-channel, cuts >3mm, no reformats, motion artifact)
* No radiology over reads by participating institution

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any participant less than 18 years old after blunt trauma
Sampling Method: Non-Probability Sample
Enrollment: 15700 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Predictive Values of CT, XR, and MRI | 5 years
  The sensitivity, specificity, negative and positive predictive values of CT, XR, and MRI for clinically significant injury will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Russell, MD, Principal Investigator — University of Utah
Locations (9):
- United States (9):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Lucile Packard Children's Hospital, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Oregon Health and Science University, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - Primary Children's Hospital, Salt Lake City, Utah